Participant Informed Consent for Clinical Research

# Study title for participants: Assessing How Normal Variations in CT Scanning Affects Its Interpretation

Official study title for internet search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Stability of Radiomic Features for Abdominal Tumors on Contrast Enhanced CT

## Lead Researcher: Kinh Gian (Richard) Do, MD, PhD at 212-639-8591

If you are the parent or legal guardian of the person who is being asked to participate in this research study, you may give consent on his or her behalf. The word "you" in this document refers to your child, if the participant is a minor, or to a person with a cognitive impairment for whom you are the Legally Authorized Representative (LAR).

## **Overview and Key Information**

## Why is this study being done?

We are asking you to take part in a clinical research study. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

Radiomics is the study on why tumors look different across patients with the same diagnosis in medical images. Therefore, the purpose of this study is to obtain additional useful pictures on your CT scan to study the tumors in a different way.

## Taking part in this study is your choice.

You can choose to take part or not to take part in this study, and you can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document presents important information to help you make your choice. Please take time to read it carefully. Talk with your doctor, family, or friends about the risks and benefits of taking part in this study. It's important that you have as much information as you need, and that all your questions are answered.

# What is the usual approach to my abdominal cancer?

You are being asked to take part in this study because you have abdominal cancer and are scheduled to have a routine Computed Tomography (CT) scan. People who are not in a study, generally have routine imaging studies done following clinical care, such as a CT scan.

## What are my other choices if I decide not to take part in this study?

- You may choose to have the usual approach described above
- You may choose to take part in a different research study, if one is available

## What will happen if I decide to take part in this study?

If you decide to take part in this study, extra pictures will be taken during the routine CT scan. Your participation in the study will be finished once the CT scan is complete.



## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important to think carefully about these as you make your decision.

#### **Risks**

We want to make sure that you know about a few key risks right now. We will also give you more information in the *What risks can I expect from taking part in this study?* section of this consent form.

There is also a risk that you could have side effects from the CT scan. These side effects may be worse, and they may be different than you would have with the usual approach for abdominal cancer.

Some of the most common side effects that the study doctors know about are:

Risks of radiation exposure

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

You will not directly benefit from the research. The research is voluntary, and you may withdraw at any time without any compromise to your routine care. The research is not a treatment and thus no treatment alternatives exist. You will receive the results of the routine CT scan from your treating doctor. If any incidental findings are detected, it will be discussed with your doctor.

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop participating in the study at any time.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

If you decide to stop, let the study doctor know as soon as possible. It's important that you stop safely.

If you stop, you can decide whether to let the study doctor or a member of the study team continue to contact you to ask questions about your health. We will not be able to withdraw information about you that has been used or shared with others before you informed us of your decision to stop.

# Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes, and the study is no longer in your best interest
- New information becomes available, and the study is no longer in your best interest
- You do not follow the study rules
- For women who are able to have children: You become pregnant while you are in the study
- The study is stopped by the National cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or the study sponsor, MSKCC. The study sponsor is the organization that oversees the study.

It is important that you understand the information in this informed consent document before you make a decision about participating in this clinical trial. Please read, or have someone read to you, the rest of



this document. If there is anything that you don't understand, ask the study doctor or nurse for more information.

## What is the purpose of this study?

Radiomics is the study on why tumors look different across patients with the same diagnosis in medical images. A CT scan is one of the most often used methods to image abdominal tumors. You are being asked to take part in this study because you have an abdominal tumor and are scheduled to undergo a routine CT scan with contrast. Our goal is to see how measurements of tumor differences vary with slight changes in CT scan parameters

About 150 people will take part in this study.

About 75 people will take part in this study at Memorial Sloan Kettering Cancer Center (MSK).

## What are the study groups?

A computer will by chance assign you to groups in the study. This is called randomization. This is done by chance because no one knows if one study group is better or worse than the other. All participants will be randomized to one of 18 different study groups. Each study group will have a research phase in their routine CT scan, which will obtain more pictures. Each research phase has a different combination of CT scan parameters.

# What extra tests and procedures will I have if I take part in this study?

#### Before you begin the main part of the study:

The study doctor will review your medical records and the results of your exams, tests, and procedures to see if it is safe for you to take part in the study. This first part of the study is called screening. Most of the screening exams, tests, and procedures are part of the usual care that you would have if you were not in a study.

The tests and procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

An additional CT image will be obtained in your CT scan.

#### **During the study:**

#### Exams, Tests and/or Procedures

You will have a CT scan during the main study. The procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

- You will have an intravenous line (IV) inserted into one arm as part of your routine CT scan
- You will be scanned on the CT scanner the same way as any other routine CT scans. However, there is a research phase that will collect extra pictures during your routine CT scan and will last approximately less than one minute

This study is not designed to affect your treatment plan, which will be decided between you and your doctor. In the unlikely event that new findings are visible on your additional CT images, these will be communicated to your doctor



#### Will I receive the results of my research tests?

Neither you nor your doctor will receive the results of any tests done for research purposes during this study.

## What risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work, school, or at home, and you may spend more time than usual in the hospital or doctor's office
- You may be asked sensitive or private questions that you do not usually discuss

The CT scan used in this study may affect how different parts of your body work, such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood throughout the study, and he or she will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drug(s)/study approach.

Important information about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may make it difficult for you to have children.
- Some side effects may be mild. Others may be very serious and may even result in death.

Important information about how you and the study doctor can make side effects less of a problem for you:

- If you notice or feel anything different, tell the study doctor. He or she can check to see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce your side effects.

The tables below show the most common and the most serious side effects that researchers know about. There may be other side effects that the doctors do not yet know about. If important new side effects are found during this study, the study doctor will discuss them with you.

#### Possible side effects of Radiation:

#### Occasional, some may be serious

In 100 people receiving CT Scan, between 4 and 20 may have:

#### Risks of Radiation Exposure:

There are no major risks associated with this study. However, even low levels of radiation are associated with a very low, unknown risk of causing cancer later in your life. CT scans require some exposure to radiation. In this study, the exposure to radiation will be increased by approximately 25-50%. We know from scientific data that the risk of developing a cancer caused by the low dose of radiation you will receive from these scans is certainly very low, if there is any risk. You should not be pregnant or lactating while undergoing this study due to the additional exposure to radiation.



# What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

- Keep your study appointments
- Tell the study doctor about:
  - o All medications and any supplements you are taking
  - o Any side effects from these medications or supplements
  - Any doctor visits or hospital stays outside of this study
  - Whether you have been or are currently in another research study

# Is there a conflict of interest for this study?

This study is sponsored by Memorial Sloan Kettering Cancer Center (MSKCC)
The study is funded by National Institutes of Health (NIH).
No conflicts of interest have been identified for either the institution or the investigator(s) in this study.

## What are the costs of taking part in this study?

The additional CT component will be done at no charge while you take part in this study. There is no cost for taking part in this study. You will not be paid for taking part in this study.

You and/or your health plan/insurance company will have to pay for all the other costs of preventing your cancer while you are in this study. These charges include the costs of insurance co-pays and deductibles, as well as tests, procedures, or drugs that you get during the study to monitor your safety, and to prevent or manage any side effects.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it does not pay for if you take part in this clinical trial. Also find out if you need approval from your health plan before you can take part in this study.

The study doctor or nurse can help you find the right person to talk to if you are not sure which costs will be billed to you or your insurance provider.

# Will I receive payment for taking part in this study?

You will not be paid for taking part in this study.

# What happens if I am injured or hurt because I took part in this study?

You will get medical treatment if you are injured as a result of taking part in this study.

If you think that you have been injured as a result of taking part in this research study, tell the study doctor or the person in charge of the study as soon as possible. The name and telephone number of the person in charge of this research are listed on the first page of this consent form.

We will offer you treatment for research injuries that happen as a result of your taking part in this study. You and/or your health plan will be charged for this treatment. Medical services will be offered at the usual charge. You will be responsible for any costs not covered by your health plan/insurance company.

If you think that your injury was a result of medical error, you keep all your legal rights to receive payment for treating the injury, even though you are in a study.



Approval date: 22-Jun-2022

## Who will see my medical information?

Your privacy is very important to us, and the researchers will make every effort to protect it. Trained staff at Memorial Hospital may review your records, if necessary.

Access to your protected health information will be limited to those listed in the Research Authorization form, which is a part of the informed consent process.

Your information may be given out, if required by law. For example, some states require doctors to make a report to the state health board if they find that a participant in a research study has a contagious disease like tuberculosis. However, the researchers will do their best to make sure that any information about you that may be released will not identify you.

In the future, your information (data) may be de-identified, which means that your data will be assigned a unique code, and the list that links the code to your name will be stored separately from your data. Your de-identified information may be used for research that has not been described in this consent form, and they may be shared with another investigator for future research. You will not be asked if you agree to take part in future research studies.

If your information from this study is used in any reports or publications, your name and anything else that could identify you will not be used. It is possible that your de-identified information from this study will be shared with other researchers outside of MSK and may be stored in public databases. All requests for data sharing will be reviewed by the study sponsor, and if individual results are included in the data, they will not contain any identifiable information about you, such as your name, address, telephone number, or social security number. Your privacy is very important to us and we use many safety procedures to protect your privacy. However, we cannot guarantee that no one will ever be able to use your information to identify you.

The study doctors have a Certificate of Confidentiality from the National Institutes of Health for this study. This gives MSK an additional way to protect sensitive information that identifies you in your records if it is requested as part of a legal proceeding. However, MSK may still be required to share some of your medical information if required by law.

## Where can I get more information?

You may visit the NCI web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about research studies, or for general information about cancer. You may also call the NCI Cancer Information Service to get the same information at 1-800-4-CANCER (1-800-422-6237).

You can talk to the study doctor about any questions or concerns that you may have about this study, or to report side effects or injuries. You may also contact the lead researcher listed on the first page of this consent.

For questions about your rights while you are participating in this study, call the MSK Institutional Review Board (IRB) at 212-639-7592. If you have concerns, complaints, or input on research, or if you would like more information about the informed consent process, please contact the MSK Patient Representative Department at 212-639-7202.



Research Authorization for the Use and Disclosure of Protected Health Information (PHI)

## Assessing How Normal Variations in CT Scanning Affects Its Interpretation

Federal law requires Memorial Sloan Kettering Cancer Center (MSK) to protect the privacy of information that identifies you and relates to your past, present, and future medical conditions (protected health information; PHI). We are committed to protecting the privacy of your information.

If you enroll in this research study, your protected health information will be used and shared with others, as explained below. MSK must obtain your permission before using or sharing your protected health information for research purposes. This form helps to make sure that you are informed of the ways in which your information will be used or shared in the future.

Carefully read the information below before you sign this form. By signing this form, you agree to the use and disclosure of your information for this research study.

# 1. What protected health information about me will be used or shared with others during this research?

- Your medical records
- Your research records, including new health information created from study-related tests, procedures, visits, and/or questionnaires
- HIV-related information, including any information indicating that you have had an HIV-related test; or that you have HIV infection, HIV-related illness, or AIDS; or any information that could indicate that you may have been exposed to HIV. (New York State requires us to obtain your consent to use or share this information.)

# 2. Who will use or share my protected health information?

MSK will use and share your protected health information. People and offices that deal with research oversight, quality assurance, and/or billing will be able to use and share your protected health information, including:

- The study's Principal Investigator and Co-Principal Investigator(s): Dr. Kinh Gian (Richard) Do, MD, PhD; & Mithat Gonen, PhD;
- Your research team at MSK, including the participating investigators, research staff, research nurses, fellows/residents, and clerical support staff
- Any healthcare personnel who provide services to you in connection with this study
- Members and staff of MSK's Institutional Review Board (IRB) and Privacy Board (PB)
- Staff of MSK's Clinical Research Administration, which oversees clinical studies, and Clinical Research Information Technology Group, which manages research databases
- Members of MSK's Data Safety Monitoring Board/Committee and the Quality Assurance Committee



# 3. With whom outside of MSK may my protected health information be shared?

Although all reasonable efforts will be made to maintain the confidentiality of your protected health information, it may be shared with and used by the following:

- The company or organization that provides the funding for the study, National Institutes of Health (NIH).
- MSK's research collaborators, business partners, subcontractors and agent(s), in the United States or in other countries, working to conduct the study, to monitor the study, or to analyze the study information for this study or for other research about the study data analysis.
- Other research doctors and medical centers participating in this research.
- Federal and state agencies, and other domestic or foreign government bodies, if required by law and/or necessary for oversight purposes, including:
  - Office for Human Research Protections (OHRP) of the US Department of Health and Human Services (HHS)
  - US Food and Drug Administration (FDA) and other regulatory agencies responsible for oversight of research
  - National Cancer Institute (NCI)/National Institutes of Health (NIH)
- Other qualified researchers, approved by MSK, who may receive individual research results that do not identify you.

Some of the organizations that may receive your protected health information may not have to satisfy the privacy rules and requirements; they may share your information with others without your permission.

# 4. Why will my protected health information be used by or shared by MSK or others?

The main reasons for the use or sharing of your information include the following:

- To conduct the study, to monitor your health status, to measure the effects of the drug(s)/device(s)/procedure(s) being studied, and to determine the research results
- To ensure that the research meets legal and institutional requirements
- To develop new tests, procedures, and commercial products
- To enhance research databases, so that scientists can design better research studies to develop new therapies for patients and to gain a better understanding of disease
- To assist with MSK medical treatment, billing, or healthcare operations. For example, medical information produced by this research study will become part of your hospital medical record.

# 5. For how long will my protected health information be used or shared with others?

There is no set date at which your protected health information that is being used or shared for this research study will be destroyed or no longer used. The information used and created during the



A16

Memorial Sloan Kettering Cancer Center IRB Number: 17-010 A(11) Approval date: 22-Jun-2022

study may be analyzed for many years, and it is not possible to know when this analysis will be completed.

# 6. Statement of privacy rights:

- It is your right to refuse to sign this authorization form. If you do not sign this form, you will not be able to participate in this research study. However, if you do not sign, it will not affect your ongoing medical treatment or healthcare coverage.
- You have the right to withdraw your permission for MSK to use or share your protected health information. Please note that we will not be able to withdraw all the information about you that already has been used or shared with others to carry out research-related activities such as oversight, or information that is needed to ensure the quality of the study. To withdraw your permission, write to the study doctor listed on the first page of this consent form at: Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, NY 10065. If you withdraw permission for us to use or share your protected health information, you will not be able to continue to participate in this research study.
- You have the right to request access to your protected health information that is being used or shared during this research and that is related to the research or to payment for the research. However, you may access this information only after the study is completed. You may have access to your medical record at any time. To request this information, please contact the study doctor whose name and telephone number are listed on the first page of this consent form. You may also ask the study doctor to correct any study-related information about you that is wrong.

#### **Notice concerning HIV-related information**

Individuals/organizations are prohibited from sharing any HIV-related information about you without your approval, unless they are permitted to do so under federal or state law. You have a right to request the list of people who may receive or use your HIV-related information without your authorization.

If you experience discrimination because of the release or disclosure of your HIV-related information, you may contact the New York State Division of Human Rights at 888-392-3644 or the New York City Commission on Human Rights at 212-306-7500. These agencies are responsible for protecting your rights.



Memorial Sloan Kettering Cancer Center IRB Number: 17-010 A(11) Approval date: 22-Jun-2022

## Participant Informed Consent/Research Authorization for Clinical Research

## Statement of professional obtaining consent

I have fully explained this clinical research study to the participant or to his/her Legally Authorized Representative (LAR). In my judgment, and in that of the participant or his/her LAR, sufficient information, including risks and benefits, was provided for the participant or his/her LAR to make an informed decision. The consent discussion will be documented in the participant's EMR.

Consenting professional must personally sign and date

| Consenting professiona signature | al's | | Date: |
|---|---|---|---|
| Consenting professiona<br>(Print) | al's name | | |
| I have read this form that described with the consenting profession this clinical research study; (2) information (data about myself of this consent form. | ribes the clin<br>al. By signing<br>to authorize<br>I/the participa | Representative's [LAR's)]) stated ical research study. I have also talked below, I agree to the following: (1) the use and disclosure of my/the pant); and (3) to state that I have received. | ed it over to my satisfaction<br>to voluntarily participate in<br>rticipant's protected health<br>ved a signed and dated copy |
| Participant/LAR must personally sign and date | | | |
| Participant/LAR | | $oxed{\mathbf{D}}$ | Pate: |
| signature Participant/LAR | | | |
| name (Print) | | | |
| LAR relationship to | | | |
| participant | | | |
| T F | <u> </u> | | |
| Witness signature (if re | quired) | | |
| participant's (or LAR's) land for the participant (or LAR) Other: I confirm that the confirmation that the confirmation that | guage, and I<br>onsent discus | sipant: I declare that I am fluent in bo<br>confirm that the consent discussion<br>sion occurred, and that the participa<br>his/her mark, or verbally agreeing. | was appropriately interpreted |
| Name of witness: | | | |
| Signature of witness: (The name of the witness must be documented in the EMR.) | | nted in the EMR.) | Date: |
| Interpreter (if required | | , | |
| Name of interpreter (if present): | | | |
| ID number (if phone interpreter): | | | |
| (The interpreter's name or ID number must be documented in the EMR.) | | | |
| The participant/Legally Aut | norized Repr | esentative must be provided with a | signed copy of this form |

